CLINICAL TRIAL: NCT06426979
Title: Sequential Letrozole and Methotrexate Therapy Safely Improved the Outcomes of Medical Treatment of Tubal Ectopic Pregnancy
Brief Title: Sequential Letrozole and Methotrexate Therapy Role in Treatment of Tubal Ectopic Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Walid Mohamed Elnagar, Assistant professor of Gynecology, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ZU-IRB#254 24/3-2024
Record Dates: First submitted 2024-05-19; First posted 2024-05-23 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Pregnancy Tubal
MeSH Terms: conditions — Pregnancy, Tubal | interventions — Methotrexate; Letrozole

STUDY DESIGN:
Who Masked: Participant
Masking Description: Patients were divided into 2 Groups as the group titles were printed into cards that were enclosed in sealed envelopes and patients were asked to choose a closed envelop.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group LTZ-MTX (Active Comparator): Letrozole and Methotrexate Therapy's Group
  Interventions: Drug: Methotrexate; Drug: Letrozole
- Group MTX (Active Comparator): Methotrexate Therapy's Group
  Interventions: Drug: Methotrexate

INTERVENTIONS:
Drug: Methotrexate — Methotrexate 25 mg/ml was given as single-dose of intramuscular (IM) injection in a dose of 50 mg/m2.
Drug: Letrozole — FEMARA 2.5 mg tablets two tablets daily
  Arms: Group LTZ-MTX

SUMMARY:
Ectopic pregnancy (EP) is a common condition involving the implantation of fertilized ovum outside the uterine cavity, accounting for 1-2% of all pregnancies. Tubal EP (TEP) is the most common and poses a significant risk to maternal life. Early diagnosis and medical treatment, such as methotrexate (MTX) and the Fallopian tube (FT), have been studied. However, the efficacy of single-dose methotrexate (SD-MTX) is questionable, and the efficacy of two-dose versus SD-MTX for medical management of EP is being evaluated. High estrogens/progesterone ratios can disrupt embryonic motility and lead to TEP.

ELIGIBILITY:
Inclusion Criteria:

* Presence of gestational masses of <3.5 cm in its greatest diameter in an intact uterine tube and showed no fetal cardiac activity;
* Absence of hemodynamic manifestations or evidence of intra-peritoneal bleeding on TVU and pre-treatment serum hCG of <3500 IU/L.

Exclusion Criteria:

* Free of Inclusion Criteria

Ages: 22 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
The Rate of resolution of Tubal Ectopic Pregnancy (TEP) | 9 months
  Role of Letrozole in resolution of Tubal Ectopic Pregnancy (TEP) that was confirmed by TVU and without shifting to surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Zagazig university, Zagazig, Ash Sharqia Governorate, Egypt